CLINICAL TRIAL: NCT04239352
Title: Levels of Inflammatory and Cardiovascular Risk Markers in Preeclamptic Patients; New Biomarkers: Pentraxin 3 & Lipoprotein-associated Phospholipase A2
Brief Title: Preeclamptic Patients and Pentraxin 3 & Lipoprotein-associated Phospholipase A2
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, Pınar kadirogullari, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ATADEK-2020/01
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Pre-Eclampsia
Keywords: Pentraxin 3; Lipoprotein-associated phospholipase A2; preeclampsia; risk markers
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pregnant women: Blood samples taken from 40 healthy pregnant women will be obtained by taking patient consent forms and storing their serum at -80 degrees. Then, serum Pentraxin 3 and Lp-PLA2 levels will be checked in these blood by ELISA method.
  this group will be the control group.
  Interventions: Diagnostic Test: Pentraxin 3 ; new biomarker; Diagnostic Test: Lipoprotein-associated phospholipase A2 ; new biomarker
- preeclamptic pregnant women: Blood samples taken from 40 preeclamptic pregnant women will be obtained by taking patient consent forms and storing their serum at -80 degrees. Then, serum Pentraxin 3 and Lp-PLA2 levels will be checked in these blood by ELISA method.
  this group will be the study group.
  Interventions: Diagnostic Test: Pentraxin 3 ; new biomarker; Diagnostic Test: Lipoprotein-associated phospholipase A2 ; new biomarker

INTERVENTIONS:
Diagnostic Test: Pentraxin 3 ; new biomarker — Pentraxin (PTX3) is an inflammatory molecule that belongs to a recently identified, well-known C-reactive protein (CRP) family.
  PTX3 plasma levels increase in vascular disorders including myocardial infarction and correlate with small vessel vasculitis and outcome or disease activity.
  These biological and clinical features of PTX3 have led us to investigate this molecule in preeclampsia, a syndrome characterized by a prominent vascular component.
Diagnostic Test: Lipoprotein-associated phospholipase A2 ; new biomarker — Lp-PLA2 is a recently described and potentially useful plasma biomarker associated with cardiovascular diseases. Because of this effect, we will investigate that preeclampsia also be beneficial.

SUMMARY:
In particular, pentraxine 3 (PTX3) molecule was assumed to have a prognostic value in acute myocardial infarction.In patients affected by acute myocardial infarction, early plasma elevation of PTX3 appears to predict a worse outcome in these patients in the longer term.

The inflammatory basis of preeclampsia resembles an atherogenic process.It is planned to investigate the role of these two molecules in endothelial dysfunction typical of preeclampsia.

The level of circulating PTX3 and Lp-PLA2 in preeclamptic patients and their serum levels according to the severity of preeclampsia and presence of IUGR, and comparison with the control group without preeclampsia and It is planned to investigate the cut-off values and sensitivity and specificity of both molecules together and separately in preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women diagnosed with preeclampsia; The blood pressure and proteinuria (at least ≥ 300 mg in urine for 24 hours) will be established before the 20th week of gestation in normotensive pregnancies with an interval of 6 hours.
* Those who have Grand mal convulsions; other causes of convulsions and exclusion of coma were defined as having seizures for the first time after 20 weeks of gestation and 48-72 hours after delivery.
* The diagnosis of HELLP syndrome will be confirmed by intravascular hemolysis. (Abnormal peripheral smear and / or abnormal bilirubin values), high liver enzymes (high serum aspartate transaminase levels [AST], alanine transferase [ALT] and lactate dehydrogenase [LDH] üst 2 upper level) and low platelet count (<100 000 / mm3)
* healthy pregnant women without additional disease for the control group

Exclusion Criteria:

* Maternal diabetes
* Kidney disease
* Cardiovascular disease
* Neurological disease
* drug use history
* Hematological and immunological disease
* The presence of any infection
* Fetal anomaly
* In utero dead fetus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: blood from 40 healthy pregnant women, 40 preeclamptic pregnant women; Serums will be stored at -80 degrees. Then, serum Pentraxin 3 and Lp-PLA2 levels will be examined in these blood by ELISA method.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
study group | 1 week
  preeclampsia in pregnant women; in the study group; serum Pentraxin 3 & Lipoprotein-associated phospholipase A levels
  It will be investigated whether these parameters observed in pregnant women with preeclampsia vary. Thus, it will be tried to be shown that these new markers may have a place in predicting the risk of preeclampsia
control group | 1 week
  in healthy pregnant women; in the control group; serum Pentraxin 3 & Lipoprotein-associated phospholipase A levels
  The values of these new parameters in healthy pregnants that constitute the control group will be determined and it will be understood whether there is a difference with the pregnants who developed the preeclampsia

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)